CLINICAL TRIAL: NCT01213095
Title: R-CVP Followed by Rituximab Maintenance Therapy for Patients With Advanced Marginal Zone B-cell Lymphoma
Brief Title: Rituximab Maintenance Therapy for Marginal Zone B-cell Lymphoma (MZL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A University Hospital (Other)
Responsible Party: Principal Investigator, Sung Yong Oh, Department of internal medicine, Dong-A University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISL-MZL-10-4(ML25403)
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2014-11

CONDITIONS: Lymphoma
Keywords: Lymphoma; B-Cell; Marginal Zone; Rituximab
MeSH Terms: conditions — Lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental): rituximab 375mg/m2, every 8 weeks, 12 times
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — rituximab 375mg/m2, every 8 weeks, 12 times

SUMMARY:
The clinical efficacy of rituximab, a chimeric monoclonal antibody targeted toward the B-cell specific antigen CD20, was initially demonstrated in cases of follicular lymphoma (FL), but the use of this antibody has been extended over the last few years to the majority of subtypes of B-cell CD20 positive non-Hodgkin's lymphomas, with promising results thus far. In MZL, small numbers of case reports have chronicled the use of rituximab as a single agent or phase II trial combination with chemotherapeutic regimens.

The results of the rituximab maintenance phase III trial demonstrated that patients with FL who continued to take rituximab monotherapy as a maintenance therapy after responding to an initial course of chemotherapy combined with or without rituximab experienced longer progression-free survival durations than did those who received no rituximab maintenance therapy. The efficacy of maintenance treatment after first-line induction treatment with R-chemotherapy was addressed in the international PRIMA (Primary Rituximab and Maintenance) study, which has enrolled 1,217 patients. The first results are eagerly awaited. Although MZL has better prognosis in TTP and OS than FL, both of them are classified as the same category of indolent lymphoma -characterized by frequent relapse and prolonged survival.

According to the results of our survey, advanced stage MZL tends to be an indolent disease - characterized by prolonged survival with frequent relapses. Rituximab appears to contribute to better responses, but not in TTP. Thus, we should consider maintenance treatments for MZL patients, to extend their response duration.

DETAILED DESCRIPTION:
no desire description

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20 positive marginal zone B-cell lymphomas
* Ann Arbor stage III or IV
* No prior chemotherapy or radiotherapy for advanced stage MZL
* Tumor response after 8th cycles of R-CVP CTx ≥ SD (Stable disease)
* Performance status (ECOG) ≤ 2
* age ≥ 20
* At least one or more bidimensionally measurable lesion(s): ≥ 2 cm by conventional CT/ ≥ 1 cm by spiral CT/ skin lesion (photographs should be taken) ≥ 2 cm/ measurable lesion by physical examination ≥ 2 cm
* Adequate renal function: serum creatinine level < 2 mg/dL (177 μmol/L)
* Adequate liver functions: Transaminase (AST/ALT) < 3 X upper normal value / Bilirubin < 1.5 X upper normal value /Alkaline phosphatase < 5 X upper normal value
* Adequate BM functions:ANC > 1500/uL and platelet > 75,000/uL and Hemoglobin > 9.0 g/dL unless abnormalities are due to bone marrow involvement by lymphoma
* Informed consent

Exclusion Criteria:

* Other subtypes NHL than MZL
* Large cell component >10%
* Tumor response after 8th cycles CTx = PD (Progression disease)
* Central nervous system (CNS) metastasis
* Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions i. Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry ii. History of significant neurologic or psychiatric disorders including dementia or seizures iii. Active uncontrolled infection (viral, bacterial or fungal infection) iv. Other serious medical illnesses
* Known hypersensitivity to any of the study drugs or its ingredients (i.e., hypersensitivity to Polysorbate 20, CHO cell products, or recombinant human antibodies)
* Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
3 year progression free survival | 3 years after last patient enrollment
  Historic 3 year progression free survival rate was 60 %, expected difference 20%, power 0.80, significance 0.05 and drop rate=0.1.

SECONDARY OUTCOMES:
Overall survival | 5 years after last patients enrollment
toxicity | during the Rituximab maintenance treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Oh, M.D., Study Director — Dong-A University Hospital
Locations (1):
- Sung Yong Oh, Busan, South Korea

REFERENCES:
- [Derived] Oh SY, Kim WS, Kim JS, Kim SJ, Yoon DH, Yang DH, Lee WS, Kim HJ, Yhim HY, Jeong SH, Won JH, Lee S, Kong JH, Lim SN, Ji JH, Kwon KA, Lee GW, Lee JH, Lee HS, Shin HJ, Suh C. Phase II study of R-CVP followed by rituximab maintenance therapy for patients with advanced marginal zone lymphoma: consortium for improving survival of lymphoma (CISL) study. Cancer Commun (Lond). 2019 Oct 16;39(1):58. doi: 10.1186/s40880-019-0403-7. PMID 31619290